CLINICAL TRIAL: NCT00556972
Title: A Feasibility Study of a Fecal Incontinence Management System for Medical Use
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to numerous delays in study start-up process...
Sponsor: Coloplast A/S (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: DK172OS
Record Dates: First submitted 2007-11-09; First posted 2007-11-12 (Estimated); Results first posted 2013-01-01 (Estimated); Last update posted 2022-12-06 (Actual); Status verified 2022-11

CONDITIONS: Fecal Incontinence
MeSH Terms: conditions — Fecal Incontinence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Fecal Incontinence management system (Experimental): Fecal Incontinence Management System is based on the same principle as fecal pouches. A barrier around anus to ensure adhesion and prevent leakage.
  Interventions: Device: Fecal Incontinence Management System

INTERVENTIONS:
Device: Fecal Incontinence Management System — The device is intended to remedy fecal incontinence.

SUMMARY:
The purpose of this feasibility study is to evaluate the performance and skin-friendliness of the barrier of the Fecal Incontinence Management System. The investigator will complete a questionnaire for each of the tested products and the products will be evaluated as regards leakage, wear time, and skin-friendliness.

DETAILED DESCRIPTION:
The purpose of this feasibility study is to evaluate the performance and skin-friendliness of the barrier of the Fecal Incontinence Management System. The investigator will complete a questionnaire for each of the tested products and the products will be evaluated as regards leakage, wear time, and skin-friendliness

ELIGIBILITY:
Inclusion Criteria:

* The subject is at least 18 years of age
* The subject has fecal incontinence

Exclusion Criteria:

* The subject is pregnant and/or breastfeeding
* The subject has perianal fistulas and/or hemorrhoids
* It's estimated that the subject's perianal skin makes it inappropriate for subject to participate in the study (i.e. in case of damaged skin, very sweaty skin or very sinuous and folded skin)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 4 (Actual)
Dates: Start 2008-01; Primary Completion 2008-04 (Actual); Study Completion 2008-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Thais Benjamin N. Christensen, M.Sc. (BME), Study Chair — Coloplast A/S
Locations (1):
- Beth Israel Deaconess Medical Center, Inc., Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Fecal Incontinence Management System: The product is a management system for use in fecal incontinence. It consists of a barrier with an attached pouch and a Bed Drainage Bag.
Period: Overall Study
Arm/Group | Fecal Incontinence Management System
Started | 4
Completed | 4
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Fecal Incontinence Management System
Number analyzed (Participants) | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 2
  >=65 years | 2
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.0 (14.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3
  Male | 1
Region of Enrollment [Number; unit: participants]
  United States | 4

OUTCOME MEASURES:

1. Primary Outcome: The Primary Outcome Measure is Device Wear Time (Time From the Device is Applied Until it is Removed)
Time Frame: 5 days
Population: ITT
Measure: Mean (Standard Deviation); unit: Hours
Arm/Group | Fecal Incontinence Management System
Number analyzed (Participants) | 4
Hours | 23.1 (0.7)

2. Secondary Outcome: Is the Barrier Size and Shape Satisfactory
Description: Percentage of subjects who answered yes to the question: is the barrier size and shape satisfactory
Time Frame: Subjects were followed for the duration of the study, an average of 23 hours
Population: ITT
Measure: Number; unit: Percentage of subjects
Arm/Group | Fecal Incontinence Management System
Number analyzed (Participants) | 4
Percentage of subjects | 100

3. Secondary Outcome: Assessment of Skin 0-2 Inches From the Edge of the Anus
Description: Skin condition scale: 1 = Normal skin without redness, 2 = Normal redness and intact skin, 3 = Abnormal redness but intact skin, 4 = Red and spotted but intact skin, 5 = Red and broken skin, 6 = Broken and bleeding skin Best skin condition score is 1, and worst skin condition score is 6.
Time Frame: Subjects were evaluated before and after test
Population: ITT
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Fecal Incontinence Management System
Number analyzed (Participants) | 4
Scores on a scale
  Before test | 2.25 (1.89297)
  After test | 3.25 (2.62996)

4. Secondary Outcome: What is Your Assessment of the Ease of Correct Application of the Anal Adhesive?
Time Frame: After application of product
Measure: Number; unit: Pouche and Bag
Units Other Than Participants: Pouch and bag
Arm/Group | Fecal Incontinence Management System
Number analyzed (Participants) | 4
Number analyzed (Pouch and bag) | 7
Pouche and Bag
  Very difficult | 0
  Difficult | 1
  Reasonable | 0
  Easy | 6
  Very Easy | 0

ADVERSE EVENTS:
Arm/Group | Fecal Incontinence Management System
Serious Adverse Events (participants affected / at risk) | 0/4
Other Adverse Events (participants affected / at risk) | 0/4

LIMITATIONS AND CAVEATS:
No overall conclusions could be drawn, due to the limited amount of data (N=4 due to delays and low recruitment rate). A new study, with a higher sample size needs to be executed, if the objectives set in this study are to be investigated thoroughly.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less